CLINICAL TRIAL: NCT03649113
Title: Percutaneous Sclerotherapy of Symptomatic Liver Hemangioma With Bleomycin
Acronym: Hemangioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Liver Hemangioma Sclerotherapy
Record Dates: First submitted 2018-07-19; First posted 2018-08-28 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2019-10

CONDITIONS: Hemangioma Liver

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm investigating the safety and efficacy of percutaneous sclerotherapy of hepatic hemangiomas with the mixture of Bleomycin and Lipiodol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sclerotherapy arm (Experimental): Patients with symptomatic liver hemangioma undergoing sclerotherapy (percutaneous injection) with 45 units of Bleomycin once during the procedure
  Interventions: Procedure: sclerotherapy arm

INTERVENTIONS:
Procedure: sclerotherapy arm — The liver mass will be punctured under guidance of ultrasonography with a 20- or 22-gauge Chiba needle. Contrast medium will be injected under fluoroscopy guidance to assess any possible communication with the biliary tree and to evaluate the amount of sclerosing agent which could be safely injected. Then, the mixture of Bleomycin (Bleocin-S; Korea United Pharm Inc., South Korea) and Lipiodol (Ultra-Fluid, Guerbet, France) will be slowly injected under continuous guidance of fluoroscopy. No more than 45 units of Bleomycin and 15 cc of Lipiodol will be injected in a single session.

SUMMARY:
Percutaneous sclerotherapy is currently a widely used treatment for subcutaneous low-flow vascular malformations. Considered as a low-flow vascular malformation, symptomatic liver hemangiomas could also theoretically be safely and effectively treated by percutaneous sclerotherapy with a mixture of Bleomycin and Lipiodol. The safety and efficacy of percutaneous sclerotherapy was firstly introduced by the investigator's investigators in 5 patients in a pilot study. The aim of this study is to design and conduct a study to evaluate the safety and efficacy of percutaneous sclerotherapy in a larger sample size with a long term follow-up.

DETAILED DESCRIPTION:
Twenty-five patients with symptomatic liver hemangioma will be enrolled after an informed consent being obtained. Patients' symptoms related to liver mass, including the pain severity being measured by visual analogue scale, discomfort, early satiety, or nausea will be recorded. Liver function tests, coagulation tests, and complete blood count will be checked before the intervention. A triple phase abdominal CT scan with the administration of intravenous contrast medium will also be performed before the procedure. Exclusion criteria include hepatic or renal impairment, abdominal symptoms unrelated to a liver mass, uncorrectable coagulopathy, lung fibrosis, allergy to contrast media, systemic infection, liver abscess, and biliary obstruction.

Patients will be sufficiently hydrated with normal saline before the procedure. Corticosteroid and prophylactic antibiotics will be administered before the procedure. Antibiotics will be continued for 3 days after the procedure.

The liver mass will be punctured under guidance of ultrasonography with a 20- or 22-gauge Chiba needle. Contrast medium will be injected under fluoroscopy guidance to assess any possible communication with the biliary tree and to evaluate the amount of sclerosing agent which could be safely injected. Then, the mixture of Bleomycin (Bleocin-S; Korea United Pharm Inc., South Korea) and Lipiodol (Ultra-Fluid, Guerbet, France) will be slowly injected under continuous guidance of fluoroscopy. No more than 45 units of Bleomycin and 15 cc of Lipiodol will be injected in a single session.

Any complication taking place during and within 30 days after the procedure will be recorded. Liver function tests, coagulation tests, and complete blood count will be repeated the day after the procedure, and 6 months after the procedure. Also, a triple phase abdominal CT scan will be repeated in 6 months, and 12 months after the intervention. The patients' symptoms will be asked by phone after 12 months. The changes in lesion size on CT scan and in patients' symptoms will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic liver hemangioma

Exclusion Criteria:

* hepatic or renal impairment
* abdominal symptoms unrelated to a liver mass
* uncorrectable coagulopathy
* lung fibrosis
* allergy to contrast media
* systemic infection
* liver abscess
* biliary obstruction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in patient satisfaction assessed by the Visual Analog Scale (VAS) after 6 months | 6 months
  Pain is subjectively assessed based on a visual analog scale (VAS) before and 6 months after intervention. Change in VAS is recorded.
  VAS is between zero (no pain at all) and 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Incidence of major adverse events | During the procedure and within 30 days after the procedure
  Incidence of major adverse events that may cause any of the following: A) Require therapy, minor hospitalization (less than 48 hours) B) Require major therapy, unplanned increase in level of care, prolonged hospitalization (more than 48 hours) C) Permanent adverse sequel D) Death
Change in hemangioma size | 6 months
  The size of the hemangioma is assessed on CT scans performed before and 6 months after the procedure. The largest diameter of the hemangioma is measured on axial images.

CONTACTS AND LOCATIONS:
Overall Officials: Hadi Rokni Yazdi, MD, Study Chair — Tehran University of Medical Sciences, Tehran, Iran
Locations (1):
- Imam Khomeini Hospital Complex, Tehran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayoobi Yazdi N, Dashti H, Batavani N, Borhani A, Shakiba M, Rokni Yazdi H. Percutaneous Sclerotherapy for Giant Symptomatic Liver Hemangiomas: A Pilot Study. J Vasc Interv Radiol. 2018 Feb;29(2):233-236. doi: 10.1016/j.jvir.2017.10.009. PMID 29414196
- [Background] van der Vleuten CJ, Kater A, Wijnen MH, Schultze Kool LJ, Rovers MM. Effectiveness of sclerotherapy, surgery, and laser therapy in patients with venous malformations: a systematic review. Cardiovasc Intervent Radiol. 2014 Aug;37(4):977-89. doi: 10.1007/s00270-013-0764-2. Epub 2013 Nov 7. PMID 24196269
- [Background] Negrier C, Delmas MC, Ranchin B, Cochat P, Dechavanne M. Decreased factor XII activity in a child with nephrotic syndrome and thromboembolic complications. Thromb Haemost. 1991 Oct 1;66(4):512-3. No abstract available. PMID 1796406
- [Background] Blaise S, Charavin-Cocuzza M, Riom H, Brix M, Seinturier C, Diamand JM, Gachet G, Carpentier PH. Treatment of low-flow vascular malformations by ultrasound-guided sclerotherapy with polidocanol foam: 24 cases and literature review. Eur J Vasc Endovasc Surg. 2011 Mar;41(3):412-7. doi: 10.1016/j.ejvs.2010.10.009. Epub 2010 Dec 15. PMID 21111641
- [Background] Mathur NN, Rana I, Bothra R, Dhawan R, Kathuria G, Pradhan T. Bleomycin sclerotherapy in congenital lymphatic and vascular malformations of head and neck. Int J Pediatr Otorhinolaryngol. 2005 Jan;69(1):75-80. doi: 10.1016/j.ijporl.2004.08.008. PMID 15627451
- [Background] Vilgrain V, Boulos L, Vullierme MP, Denys A, Terris B, Menu Y. Imaging of atypical hemangiomas of the liver with pathologic correlation. Radiographics. 2000 Mar-Apr;20(2):379-97. doi: 10.1148/radiographics.20.2.g00mc01379. PMID 10715338